CLINICAL TRIAL: NCT05676957
Title: A Prospective, Randomized-controlled Trial to Assess the Safety and Efficacy of Intravascular Hypothermia in Acute Ischemia Stroke Patients With Recanalization After Thrombectomy
Brief Title: Reperfusion With Hypothermia in Acute Ischemic Stroke
Acronym: RESCUE-HYPO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Liping Liu (Other)
Responsible Party: Sponsor-Investigator, Liping Liu, Professor, Beijing Tiantan Hospital
Organization: Beijing Tiantan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RESCUE-HYPO
Record Dates: First submitted 2023-01-03; First posted 2023-01-09 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Ischemic Stroke; Revascularization; Endovascular Treatment; Reperfusion Injury
Keywords: Ischemic Stroke; Revascularization; Endovascular Treatment; Reperfusion Injury
MeSH Terms: conditions — Ischemic Stroke; Reperfusion Injury

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): The subjects will be considered to be enrolled in the study group of the trial when all inclusion and exclusion criteria have been met, the informed consent form has been signed, and randomization to the study group of the trial to allow endovascular therapy with the Thermogard XP3 Intravascular Temperature Management (IVTM) System after recanalization.
  Interventions: Device: Thermogard XP3
- Control group (No Intervention): The subjects will be considered to be enrolled in the control group of the trial when all inclusion and exclusion criteria have been met, the informed consent form has been signed, and randomization to the control group of the trial.

INTERVENTIONS:
Device: Thermogard XP3 — Patients received endovascular hypothermia for 12 hours following endovascular treatment and recanalization.
  Other Names: intravascular hypothermia treatment
  Arms: Study group

SUMMARY:
The primary objective of this study is to determine the feasibility and safety of receiving intravascular hypothermia treatment for patients experiencing endovascular treatment after acute ischemic stroke(AIS) due to a large vessel occlusion.

DETAILED DESCRIPTION:
Hypothermia has been confirmed and widely applied in the treatment of coma patients after resuscitation from cardiac arrest, but its effect on the prognosis of patients with AIS is still controversial. Previous basic research has confirmed that hypothermia can significantly reduce the infarct volume and improve the survival rate and behavioral defects of mice by protecting ischemic brain tissue and improving reperfusion injury through a variety of ways. Therefore, we hypothesized that hypothermia can improve the prognosis of patients with AIS after reperfusion by improving reperfusion injury. This is a phase II clinical trial to to verify the efficacy and safety of endovascular hypothermia in these patients,This study enrolled patients with massive cerebral infarction after endovascular treatment recanalization, patients are divided into study group and control group. The study group received endovascular hypothermia for 12 hours following endovascular treatment and recanalization, and the control group received only usual medical treatment following endovascular treatment and recanalization. We will preliminarily explore the mechanism of endovascular hypothermia in successful reperfusion of large vessel occlusion AIS, and to provide reference for the design of future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-80 years;
* Patients with symptoms consistent with an AIS;
* Pre-stroke mRS score 0-1;
* NIHSS score 6-30 at the time of randomization;
* Computed Tomography Angiography (CTA) or Magnetic Resonance Angiography(MRA) proved occlusion of Internal Carotid Artery (ICA) terminal or M1 segment of Middle Cerebral Artery;
* Imaging showed massive infarction: within 24h of onset and Alberta Stroke Program Early CT Score (ASPECTS) < 3, and large infarct core 70-100 ml (CT perfusion [ Relative Cerebral Blood Flow (rCBF) < 30%]); within 24h of onset and ASPCECTS score 3-5 (based on NCCT); ASPECTS > 5, within 6h-24h of onset,and large infarct core 70-100 ml (CTP [rCBF < 30%]);
* Successful recanalization of occluded vessel (modified Thrombolysis in Cerebral Infarction (mTICI) scores 2b/3) after EVT;
* Patients and/or their families agreed to enter the trial.

Exclusion Criteria:

* CT after reperfusion showed PH2 hemorrhagic transformation;
* bilateral stroke or multiple intracranial occlusions;
* known presence of Inferior Vena Cava (IVC) filter;
* end-stage renal disease on hemodialysis;
* known hemorrhagic diathesis, coagulation factor deficiency or platelet count < 5 × 109/L, International Normalized Ratio(INR) > 1.7;
* known hypersensitivity to meperidine, buspirone, midazolam and other sedative and analgesic drugs;
* pregnant women;
* combined malignant tumors, sepsis, hypothyroidism;
* unstable vital signs/dying state, requiring vasoactive drugs to maintain hemodynamic stability and in the incremental phase;
* cardiac function grade 4/severe liver and kidney dysfunction;
* has participated in other drugs or device clinical trials that may have an impact on the current study;
* other reasons lead the investigator to believe that patients are not suitable to continue hypothermia treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of study group patients achieving target temperature < 34 ºC within 2 hour after recanalization. | 2 hour after thrombectomy
  Percentage of study group patients achieving target temperature < 34 ºC within 2 hour after recanalization.
final infarct volume（FIV） | three to seven days after endovascular therapy
  Infarct volume was assessed according to the non-contrast Computed Tomography (NCCT) 3-7 days after surgery, and if several NCCT examinations were performed within 3-7 days, the last CT was used.

SECONDARY OUTCOMES:
the rate of 90-day modified Rankin Scale (mRS)(0-2) | 90 days
  Compare the rate of 90-day mRS (0-2) between study group and control group
The rate of early neurological deterioration | 24 hours
  increasing of National Institute of Health Stroke Scale(NIHSS) ≥ 4 points 24 hours after recanalization
The rate of mortality | 90 days
  The rate of mortality
Systematic Intracranial Hemorrhagr(sICH) | 24 ±3hours
  sICH with 24 ±3h post recanalization

CONTACTS AND LOCATIONS:
Overall Officials: Liping Liu, Principal Investigator — Beijing Tiantan Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Powers WJ, Rabinstein AA, Ackerson T, Adeoye OM, Bambakidis NC, Becker K, Biller J, Brown M, Demaerschalk BM, Hoh B, Jauch EC, Kidwell CS, Leslie-Mazwi TM, Ovbiagele B, Scott PA, Sheth KN, Southerland AM, Summers DV, Tirschwell DL. Guidelines for the Early Management of Patients With Acute Ischemic Stroke: 2019 Update to the 2018 Guidelines for the Early Management of Acute Ischemic Stroke: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2019 Dec;50(12):e344-e418. doi: 10.1161/STR.0000000000000211. Epub 2019 Oct 30. PMID 31662037
- [Background] Goyal M, Menon BK, van Zwam WH, Dippel DW, Mitchell PJ, Demchuk AM, Davalos A, Majoie CB, van der Lugt A, de Miquel MA, Donnan GA, Roos YB, Bonafe A, Jahan R, Diener HC, van den Berg LA, Levy EI, Berkhemer OA, Pereira VM, Rempel J, Millan M, Davis SM, Roy D, Thornton J, Roman LS, Ribo M, Beumer D, Stouch B, Brown S, Campbell BC, van Oostenbrugge RJ, Saver JL, Hill MD, Jovin TG; HERMES collaborators. Endovascular thrombectomy after large-vessel ischaemic stroke: a meta-analysis of individual patient data from five randomised trials. Lancet. 2016 Apr 23;387(10029):1723-31. doi: 10.1016/S0140-6736(16)00163-X. Epub 2016 Feb 18. PMID 26898852
- [Background] Hypothermia after Cardiac Arrest Study Group. Mild therapeutic hypothermia to improve the neurologic outcome after cardiac arrest. N Engl J Med. 2002 Feb 21;346(8):549-56. doi: 10.1056/NEJMoa012689. PMID 11856793
- [Background] Hui J, Feng J, Tu Y, Zhang W, Zhong C, Liu M, Wang Y, Long L, Chen L, Liu J, Mou C, Qiu B, Huang X, Huang Q, Zhang N, Yang X, Yang C, Li L, Ma R, Wu X, Lei J, Jiang Y, Liu L, Gao G, Jiang J; LTH-1 Trial collaborators. Safety and efficacy of long-term mild hypothermia for severe traumatic brain injury with refractory intracranial hypertension (LTH-1): A multicenter randomized controlled trial. EClinicalMedicine. 2021 Jan 28;32:100732. doi: 10.1016/j.eclinm.2021.100732. eCollection 2021 Feb. PMID 33681741
- [Background] Liu X, Wen S, Zhao S, Yan F, Zhao S, Wu D, Ji X. Mild Therapeutic Hypothermia Protects the Brain from Ischemia/Reperfusion Injury through Upregulation of iASPP. Aging Dis. 2018 Jun 1;9(3):401-411. doi: 10.14336/AD.2017.0703. eCollection 2018 Jun. PMID 29896428
- [Background] van der Worp HB, Sena ES, Donnan GA, Howells DW, Macleod MR. Hypothermia in animal models of acute ischaemic stroke: a systematic review and meta-analysis. Brain. 2007 Dec;130(Pt 12):3063-74. doi: 10.1093/brain/awm083. Epub 2007 May 3. PMID 17478443
- [Background] Su Y, Fan L, Zhang Y, Zhang Y, Ye H, Gao D, Chen W, Liu G. Improved Neurological Outcome With Mild Hypothermia in Surviving Patients With Massive Cerebral Hemispheric Infarction. Stroke. 2016 Feb;47(2):457-63. doi: 10.1161/STROKEAHA.115.009789. Epub 2015 Dec 22. PMID 26696645
- [Background] Hemmen TM, Raman R, Guluma KZ, Meyer BC, Gomes JA, Cruz-Flores S, Wijman CA, Rapp KS, Grotta JC, Lyden PD; ICTuS-L Investigators. Intravenous thrombolysis plus hypothermia for acute treatment of ischemic stroke (ICTuS-L): final results. Stroke. 2010 Oct;41(10):2265-70. doi: 10.1161/STROKEAHA.110.592295. Epub 2010 Aug 19. PMID 20724711
- [Background] Lyden P, Hemmen T, Grotta J, Rapp K, Ernstrom K, Rzesiewicz T, Parker S, Concha M, Hussain S, Agarwal S, Meyer B, Jurf J, Altafullah I, Raman R; Collaborators. Results of the ICTuS 2 Trial (Intravascular Cooling in the Treatment of Stroke 2). Stroke. 2016 Dec;47(12):2888-2895. doi: 10.1161/STROKEAHA.116.014200. Epub 2016 Nov 10. PMID 27834742
- [Background] Eltzschig HK, Eckle T. Ischemia and reperfusion--from mechanism to translation. Nat Med. 2011 Nov 7;17(11):1391-401. doi: 10.1038/nm.2507. PMID 22064429
- [Background] Wu C, Zhao W, An H, Wu L, Chen J, Hussain M, Ding Y, Li C, Wei W, Duan J, Wang C, Yang Q, Wu D, Liu L, Ji X. Safety, feasibility, and potential efficacy of intraarterial selective cooling infusion for stroke patients treated with mechanical thrombectomy. J Cereb Blood Flow Metab. 2018 Dec;38(12):2251-2260. doi: 10.1177/0271678X18790139. Epub 2018 Jul 18. PMID 30019993
- [Background] Horn CM, Sun CH, Nogueira RG, Patel VN, Krishnan A, Glenn BA, Belagaje SR, Thomas TT, Anderson AM, Frankel MR, Schindler KM, Gupta R. Endovascular Reperfusion and Cooling in Cerebral Acute Ischemia (ReCCLAIM I). J Neurointerv Surg. 2014 Mar;6(2):91-5. doi: 10.1136/neurintsurg-2013-010656. Epub 2013 Mar 6. PMID 23468538
- [Background] Hong JM, Lee JS, Song HJ, Jeong HS, Choi HA, Lee K. Therapeutic hypothermia after recanalization in patients with acute ischemic stroke. Stroke. 2014 Jan;45(1):134-40. doi: 10.1161/STROKEAHA.113.003143. Epub 2013 Nov 7. PMID 24203846